CLINICAL TRIAL: NCT06007313
Title: A Cross-sectional Study of the Relationship Between Mental Stress and Bowel Preparation
Brief Title: Mental Stress and Bowel Preparation Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: swyclinical2023
Record Dates: First submitted 2023-08-07; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Colonoscopy; Intestinal Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional study was to explore the relationship between physical and psychological stress and the quality of bowel preparation before a colonoscopy examination, in order to improve the quality of bowel preparation.

The main questions it aims to answer are:

Does physical and psychological stress affect the quality of colonoscopic bowel preparation, and delay disease detection? How can we improve the quality of colonoscopy？ Participants will be asked to complete a questionnaire containing their demographics, history of diseases and drugs, lifestyle habits, and physical and 14-item perceived stress scale(PSS-14). Quality of bowel preparation was assessed by the Boston bowel preparation scale（BPS）.

DETAILED DESCRIPTION:
A total of 1000 patients who were to undergo colonoscopy at the Endoscopy Centre of the Department of Gastroenterology, Renji Hospital, from May 2023 to August 2023 were collected, and the general information and the physical and mental stress test scale of the patients were collected by questionnaires from random samples, and they were screened for enrolment according to the inclusion and exclusion criteria. The correlation between physical and mental stress and the quality of bowel preparation for colonoscopy was analyzed according to the Boston Rating Scale (BPS), which is used by colonoscopists to assess the quality of bowel preparation for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 75 years old with an indication for colonoscopy
* Participants signed an informed consent form for colonoscopy and underwent colonoscopy
* Participants not be with a history of digestive tumors, active inflammatory bowel disease and other conditions that significantly affect colonic motility
* Participants with good communication and comprehension skills and be able to answer assessment questions accurately

Exclusion Criteria:

* Withdrawal prior to colonoscopy
* Incomplete completion of information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent colonoscopy from May 2023-August 2023 at the Endoscopy Centre, Renji East Hospital.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
The quality of bowel preparation | During colonoscopy, about 20 minutes
  Quality of bowel preparation was assessed by the Boston bowel preparation scale(BPS). The BPS is used to assess the quality of bowel preparation on a 9-point scale. The colon is divided into three sections (right-sided colon, transverse colon and left-sided colon) and each segment is scored on a four-point scale (0-3), with higher scores indicating a cleaner bowel. The total Boston score is 9, with a score of less than 6 indicating poor bowel preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China